CLINICAL TRIAL: NCT04828187
Title: Development and Validation of Deep Neural Networks for Blinking Identification and Classification
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Associate Professor of Ophthalmology, Democritus University of Thrace
Other Study IDs: ES2/Th15/25-2-2021
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Blinking; Deep Learning
Keywords: deep learning; DeepLabv3+; iris and sclera segmentation; eye blink detection; complete and incomplete blink classification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: 8 patients aged between 18 to 75 years with Uncorrected Distance Visual Acuity ≥ 5/10
  Interventions: Diagnostic Test: Comparison of the proposed artificial network with the ground truth

INTERVENTIONS:
Diagnostic Test: Comparison of the proposed artificial network with the ground truth — Both eyes will be included for each study participant. Participants watched a 4-10-minute video in standard mesopic environmental lighting conditions at 3.5m viewing distance. Simultaneously, all blinking moves will be recorded through a web infrared camera.
  The proposed system was tested on the 8 different subjects. Several metrics of blink detection and classification accuracy were calculated against the ground truth, which was generated by 3 independent experts, whose conflicts were resolved by a senior expert. Two independent blink identifications are assumed to be in agreement, if and only if there is sufficient temporal overlapping and the type of blink is the same between the DLED system and the ground truth.

SUMMARY:
Primary objective of this study is the development and validation of a system of deep neural networks which automatically detects and classifies blinks as "complete" or "incomplete" in image sequences.

DETAILED DESCRIPTION:
This method is based on iris and sclera segmentation in both eyes from the acquired images, using state of the art deep learning encoder-decoder neural architectures (DLED). The sequence of the segmented frames is post-processed to calculate the distance between the eyelids of each eye (palpebral fissure) and the corresponding iris diameter. Theses quantities are temporally filtered and their fraction is subject to adaptive thresholding to identify blinks and determine their type, independently for each eye. The two DLEDs were trained with manually segmented images and the post-process was parameterized using a 4-minute video. After DLED training, the proposed system was tested on 8 different subjects, each one with a 4-10-minute video. Several metrics of blink detection and classification accuracy were calculated against the ground truth, which was generated by 3 independent experts, whose conflicts were resolved by a senior expert. Two independent blink identifications are assumed to be in agreement, if and only if there is sufficient temporal overlapping and the type of blink is the same between the DLED system and the ground truth.

ELIGIBILITY:
Inclusion Criteria

* Uncorrected Distance Visual Acuity above 6/12

Exclusion Criteria:

* corneal opacities
* age-related macular degeneration
* diagnosis of psychiatric diseases
* former eyelid surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged from 18 to 75 years with Uncorrected Distance Visual Acuity ≥ 5/10
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Identification of complete and incomplete blinks | up to 1 week
  Complete and incomplete blinks are defined by the "length of palpebral fissure-to-iris diameter" ratio
First frame of each blink | up to 1 week
  The frame in which the upper eyelid starts to move down and cover the cornea
Last frame of each blink | up to 1 week
  The frame in which eyelids open fully after a blink

SECONDARY OUTCOMES:
Length of palpebral fissure of both eyes | up to 1 week
  The distance between the upper eyelid margin and the lower eyelid margin (ie. the vertical dimension of the palpebral fissure),
Iris diameter of both eyes | up to 1 week
  The horizontal diameter of the iris (ie. the horizontal white-to white distance)

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, MD,PhD, Study Chair — Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupolis, Greece
Locations (2):
- Greece (2):
  - Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros
  - Department of Computer Science and Biomedical Informatics, University of Thessaly, Lamia, Thessaly

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nousias G, Panagiotopoulou EK, Delibasis K, Chaliasou AM, Tzounakou AM, Labiris G. Video-Based Eye Blink Identification and Classification. IEEE J Biomed Health Inform. 2022 Jul;26(7):3284-3293. doi: 10.1109/JBHI.2022.3153407. Epub 2022 Jul 1. PMID 35213320